CLINICAL TRIAL: NCT02156648
Title: A Feasibility Study for Women Receiving Adjuvant or Neo-adjuvant Anthracycline Chemotherapy With or Without Radiation for HER2-neu Positive Invasive Ductal Carcinoma
Brief Title: A Feasibility Study for Women Receiving Anthracycline Chemotherapy With or Without Radiation for HER2-neu Positive Invasive Ductal Carcinoma
Acronym: OTT14-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20140259-01H
Record Dates: First submitted 2014-05-12; First posted 2014-06-05 (Estimated); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: Invasive ductal; HER2-neu positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Feasibility Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Feasibility study (Other): All participants will have blood draws for biomarkers during the course of the study at visit 1, 2, 3, 4, 5, 6, 7 and 8. they will also have the speckle tracking echocardiogram at visit 1, 4, 5, 6, 7 and 8. For women 45 an over a cardiac PET scan will be performed at visit 1 and 5.
  Interventions: Other: Feasibility study

INTERVENTIONS:
Other: Feasibility study — All participants will have blood draws for biomarkers during the course of the study at visit 1, 2, 3, 4, 5, 6, 7 and 8. they will also have the speckle tracking echocardiogram at visit 1, 4, 5, 6, 7 and 8. For women 45 an over a cardiac PET scan will be performed at visit 1 and 5.

SUMMARY:
The purpose of this project is to assess the feasibility of collecting plasma samples for cardiac biomarker assessment, and to identify if there is an associations between the biomarkers, echocardiographic features and the cardiac PET scan results (in patients receiving radiation therapy). This is the first step in a research program that has an overall goal of being able to predict early-treatment induced cardiotoxicity in patients with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Stage I-III, HER2-neu positive invasive ductal carcinoma
2. Scheduled to receive adjuvant/neo-adjuvant 5-Fluorouracil, Epirubicin, Cyclophosphamide and Docetaxel (FEC-D) chemotherapy
3. Scheduled to receive adjuvant Trastuzumab
4. ECOG Performance status 0-2
5. Adequate baseline imaging on transthoracic echocardiography, and baseline cardiac ejection fraction of ≥ 55%. Additionally, breast cancer patients≥45 years of age and scheduled to receive whole breast radiation therapy will receive two cardiac PET scans.

Exclusion Criteria:

1. Prior anthracycline chemotherapy
2. History of dilated cardiomyopathy, congestive heart failure, or coronary artery disease
3. Life expectancy less than 15 months
4. Pregnant or lactating women
5. Use of beta receptor antagonists, calcium channel antagonists, angiotensin converting enzyme inhibitors, or angiotensin receptor inhibitors at baseline.
6. Previous chest wall/breast or nodal radiation.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-08; Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Recruitment rates | every 4 weeks up to 2 years

SECONDARY OUTCOMES:
Cardiotoxicity | Once when the last participant completes week 57
  To measure biomarkers, myocardial perfusion, cardiac adverse events and peak systolic longitudinal strain.

CONTACTS AND LOCATIONS:
Overall Officials: Susan Dent, Oncologist, Principal Investigator — The Ottawa Hospital Cancer Centre
Locations (1):
- The Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada